CLINICAL TRIAL: NCT04361747
Title: Effectiveness of Nursing Counseling on Stress and Depression for Women With Recurrent Miscarriage: A Randomized Controlled Pilot Study
Brief Title: Nursing Counseling on Stress and Depression for Women With Recurrent Miscarriage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chung-Hey Chen, Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOST 104-2314-B-006-048-MY3
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Care in Women With History of Recurrent Miscarriage
Keywords: recurrent miscarriage; nursing counseling; perceived stress; depression
MeSH Terms: conditions — Abortion, Habitual; Depression

STUDY DESIGN:
Intervention Model Description: During the 12-week prenatal genetic testing evaluation period, experimental-group participants received three nursing consultation sessions plus regular care, while their control-group peers received regular care only.
Who Masked: Participant
Masking Description: The 62 women who met the inclusion criteria were assigned systematically from a random starting point using a week as the unit (Yang & Chen, 2018) to either the experimental group (n = 31) or the control group (n = 31). To avoid contaminating data by allowing participants to communicate with one another during the prenatal genetic testing evaluation, data were collected on the first week from experimental-group participants, who were selected by a research assistant who draw lots (E for experimental group and C for control group) from a sack. Subsequently, the group allotment for the following week was systematically assigned in sequence to either the control group or the experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nursing counseling intervention (Experimental): The nursing counseling intervention was implemented by a maternity nursing instructor. During the 12-week prenatal genetic testing evaluation period, experimental-group participants received three nursing consultation sessions plus regular care, while their control-group peers received regular care only. The counseling intervention was designed to facilitate self-awareness, reduce self-blame, clarify doubts, listen to patient concerns, promote forward thinking, and encourage life planning.
  Interventions: Behavioral: nursing counseling
- control group (No Intervention): control group participants received regular care only

INTERVENTIONS:
Behavioral: nursing counseling — The counseling intervention was designed to facilitate self-awareness, reduce self-blame, clarify doubts, listen to patient concerns, promote forward thinking, and encourage life planning.
  Arms: nursing counseling intervention

SUMMARY:
Recurrent miscarriage is a frustrating event for couples. The purpose of this randomized, controlled trial was to examine the effectiveness of nursing counseling on sleep quality, depression, stress, and social support in women with recurrent miscarriage (RM). Sixty-two eligible women were randomly assigned to the experimental group (n = 31) or the control (n = 31) group. The experimental group received routine care and three sessions of nursing counseling during the 12-week prenatal genetic testing stage, while the control group received routine care only. Outcome measures included the Pittsburgh Sleep Quality Index, Edinburgh Prenatal Depression Scale, Perceived Stress Scale, and Interpersonal Support Evaluation List. Paired sample t-tests were conducted before and after nursing counseling to measure whether there were any statistically significant changes in outcome variables.

DETAILED DESCRIPTION:
2.1 | Design and sample A single-blind, randomized, controlled trial with a prospective pretest-posttest experimental design was used. Prospective participants were recruited from the obstetrics and gynecology clinic of a medical center in southern Taiwan. The inclusion criteria were (1) having experienced at least two consecutive miscarriages and (2) providing informed consent to participate. A convenience sample of 62 women meeting the inclusion criteria were enrolled in this study as participants.

2.2 | Intervention The nursing counseling intervention was implemented by a maternity nursing instructor. During the 12-week prenatal genetic testing evaluation period, experimental-group participants received three nursing consultation sessions plus regular care, while their control-group peers received regular care only. The counseling intervention was designed to facilitate self-awareness, reduce self-blame, clarify doubts, listen to patient concerns, promote forward thinking, and encourage life planning.

2.4 | Procedure and ethical considerations This study was conducted between October 2016 and January 2018 after approval had been obtained from the research ethics committee of the participating institution. The objectives of this study and the rights of participants were fully explained to each participant. Participation in this study was voluntary, and refusal to participate had no impact on subsequent access to or quality of care.

The 62 women who met the inclusion criteria were assigned systematically from a random starting point using a week as the unit (Yang & Chen, 2018) to either the experimental group (n = 31) or the control group (n = 31). To avoid contaminating data by allowing participants to communicate with one another during the prenatal genetic testing evaluation, data were collected on the first week from experimental-group participants, who were selected by a research assistant who draw lots (E for experimental group and C for control group) from a sack. Subsequently, the group allotment for the following week was systematically assigned in sequence to either the control group or the experimental group. All of the participants completed the Demographic Data Form, PSQI, EPDS, PSS, and ISEL questionnaires at pretest (immediately prior to the prenatal genetic testing evaluation) and at post-test (12 weeks post-intervention). The post-test set of questionnaires was mailed to all of the participants for completion and return to the researchers in the included postage-paid, pre-addressed envelope. Thirty experimental-group participants and 28 control-group participants completed both pretest and post-test questionnaires. The CONSORT flow diagram for this study is shown in Figure 1.

2.5 | Statistical analysis Data in this study were analyzed using the SPSS (version 17.0 for Windows, SPSS Inc., Chicago, IL, USA) statistical software package. Tests used to analyze differences in baseline characteristics between the two groups included the Chi-square (χ2) test for categorical variables and the t-test for continuous variables. Paired sample t-tests were conducted before and after nursing counseling to measure whether there were any statistically significant changes in outcome variables. All results with p < .05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* (1) having experienced at least two consecutive miscarriages and (2) providing informed consent to participate.

Exclusion Criteria:

-

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 12 weeks
  Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989). A PSQI global score of > 5 was adopted to indicate poor sleep quality, which yields a diagnostic sensitivity of 98.7% and specificity of 84.4% for diagnosing sleep disturbances (Backhaus et al., 2002). The summed scores for the seven components form a global PSQI score (range = 0-21); higher scores indicate poorer sleep quality.
Edinburgh Prenatal Depression Scale (EPDS) | 12 weeks
  The severity of depressive symptoms in our study participants during the previous week was measured using the EPDS (Cox, Holden, & Sagovsky, 1987). The EPDS consists of 10 items on a 4-point scale from 0 (not at all) to 3 (yes, most of the time). Total scores range from 0 to 30. Higher scores indicate more depressive symptoms. EPDS can be used as a screening tool for depression in pregnant and postnatal women, and has been shown to have good reliability (Da Costa, Larouche, Dritsa, & Brender, 2000; Eberhard-Gran, Eskild, Tambs, Opjordsmoen, & Samuelsen, 2001; Evans, Heron, Francomb, Oke, & Golding, 2001). In Taiwan, the Chinese-language version of the EPDS has good internal consistency (Heh, 2001; Hsu & Chen, 2008; Ko et al., 2010; Su et al., 2007), concurrent validity of 0.79 with the Beck Depression Inventory (Heh, 2001), and a sensitivity of 83% and specificity of 89% (Su et al., 2007). The Cronbach's alpha value for our study using the EPDS was 0.90.
Perceived Stress Scale (PSS) | 12 weeks
  The PSS was designed to measure the degree to which a person appraises the situations in one's life as stressful. Items of the PSS were designed to express how unpredictable, uncontrollable, and overloaded respondents find their lives to be (Cohen, Kamarch, & Mermelstein, 1983). The 10 items on the scale are rated by the subject on a 4-point scale representing the frequency with which each item occurred. The greater the stress, the higher the scores. The Chinese version of the PSS has adequate internal consistency, test-retest reliability, and construct validity.
Interpersonal Support Evaluation List (ISEL) | 12 weeks
  Social support was examined using the ISEL Short Form (Cohen, Mermelstein, Kamarch, & Hoberman, 1985). This scale measures four types of social support: tangible, appraisal, self-esteem, and belonging. It consists of 16 items with a 4-point scale ranging from (0) definitely false, to (3) definitely true. The higher the score, the higher the level of perceived social support is. The Chinese version of the ISEL Short Form has adequate convergent validity (r = 0.55 with the Social Support Index), internal consistency (α = 0.81), and test-retest reliability (r = 0.77) (Chen et al., 1994). Cronbach's α in the present study was 0.90.

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Lin Kuo, MD, Study Director — College of Medicine, National Cheng-Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No